CLINICAL TRIAL: NCT00755092
Title: Analgesic Efficacy of Doula in Nulliparous and Multiparous Women
Brief Title: Effect of Doula in Nulliparas and Multiparas
Acronym: DINAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing Medical University (Other)
Responsible Party: XiaoFeng Shen, Nanjing Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: NMU-FY2008-416; NJFY-MZ08092
Record Dates: First submitted 2008-09-17; First posted 2008-09-18 (Estimated); Last update posted 2009-02-11 (Estimated); Status verified 2009-02

CONDITIONS: Labor Pain
Keywords: Doula; Psychological care; Labor analgesia
MeSH Terms: conditions — Labor Pain | interventions — Doulas

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Doula for Nulliparous women
  Interventions: Behavioral: Doula
- 2 (Active Comparator): Doula for Multiparous women
  Interventions: Behavioral: Doula

INTERVENTIONS:
Behavioral: Doula — Doula support for nulliparous women from the beginning of regular contraction of uterus to the end of delivery
  Arms: 1
Behavioral: Doula — Doula support for multiparous women from the beginning of regular contraction of uterus to the end of delivery
  Arms: 2

SUMMARY:
Psychological care during labor is considered as an important supplemental procedure for alleviating delivering stress and pain. Although Doula has been recommending that should be given for parturients, its precise effect on nulliparous and multiparous women is still unknown. The investigators hypothesized that multiparas had experienced the process of labor, but the nulliparas were not, so Doula support would produce different effect on these two population.

ELIGIBILITY:
Inclusion Criteria:

* Healthy term parturients
* Chinese
* 19-45 years

Exclusion Criteria:

* Organic dysfunction
* Participants younger than 19 years or older than 45 years
* Those who were not willing to or could not finish the whole study at any time
* Pregnancy-induced hypertension and diabetes mellitus

Ages: 19 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2008-09; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
VAS pain intensity | From the beginning of regular contraction of uterus to the end of delivery

SECONDARY OUTCOMES:
Ramsey sedative scale | From the beginning of regular contraction of uterus to the end of delivery
Blood levels of corticosteroid | 10 min prior to Doula, 5, 10, 15, 30, 60, 120 min after Doula support and at the end of the delivery
Vital signs | From the beginning of regular contraction of uterus to the end of delivery
Adverse events | From the beginning of regular contraction of uterus to the end of delivery
Infant outcomes | The time of delivery to 1 h after delivery
Cesarean rate | During the whole period of laboring
Overall feeling of satisfaction of analgesia | From the beginning of regular contraction of uterus to the end of the labor

CONTACTS AND LOCATIONS:
Overall Officials: XiaoFeng Shen, MD, Principal Investigator — Nanjing Medical University
Locations (1):
- Nanjing Medical University, Nanjing, Jiangsu, China